CLINICAL TRIAL: NCT00713453
Title: Muscle Response to Enzyme Replacement Therapy in Pompe Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Yin-Hsiu Chien, M.D., PhD., National Taiwan University Hospital
Other Study IDs: 200704066R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Pompe Disease
Keywords: Pompe disease; muscle; enzyme replacement therapy
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to study the response of muscle cells from Pompe disease after enzyme replacement therapy

ELIGIBILITY:
Inclusion Criteria:

* patients with Pompe disease, prepare or on enzyme replacement therapy
* signed informed consent

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with Pompe disease, prepare or on enzyme replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2007-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
all morphology changes improvement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan